CLINICAL TRIAL: NCT02858128
Title: WHOLE-BODY DIFFUSION-WEIGHTED MAGNETIC RESONANCE IMAGING (WB-DW-MRI) VS CHOLINE-POSITRON EMISSION TOMOGRAPHY-COMPUTED TOMOGRAPHY (CHOLINE- PET/CT) for Selecting Treatments in Recurrent Prostate Cancer
Brief Title: WB-DW-MRI vs CHOLINE-PET/CT for Selecting Treatments in Recurrent Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Hospital Provincial de Castellon (Other)
Responsible Party: Principal Investigator, Antonio J Conde Moreno, MD PhD, Hospital Provincial de Castellon
Other Study IDs: PRV00024
Record Dates: First submitted 2016-08-03; First posted 2016-08-08 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: IMAGING STUDY — Choline-PET/CT versus NMRscan comparative study

SUMMARY:
The purpose of this study is to determine the effectiveness of whole-body diffusion-weighted magnetic resonance imaging (WB-DW- MRI) in detecting metastases by comparing the results with those from choline-positron emission tomography-computed tomography (choline-PET/CT) in patients with metastatic/oligometastatic prostate cancer. Patients with this disease profile who could benefit from treatment with stereotactic body radiation therapy (SBRT) were selected and their responses to these techniques were rated.

DETAILED DESCRIPTION:
This was a prospective, controlled, unicentric study, involving 46 consecutive patients from our centre who presented biochemical relapse after adjuvant, salvage or radical treatment with external beam radiotherapy, or brachytherapy. After initial tests ( bone scintigraphy, CT, pelvic MRI) 35 patients with oligometastases or without them were selected. 11 patients with multiple metastases were excluded from the study. WB-DW- MRI and choline-PET/CT was then performed on each patient within one week. The results were interpreted by specialists in nuclear medicine and MRI. If they were candidates for treatment with ablative SBRT (SABR) they were then evaluated every three months with both tests.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer histologic diagnostic after one treatment
* 5 o less lessions
* Asimptomatic lessions
* Informed Consent Form signed

Exclusion Criteria:

* Not capability to perform NMR os CT/PET scans

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 46 consecutive patients given a diagnosis of prostate cancer by the Radiation Oncology Department of our center, between October 2014 and March 2015 who met the established inclusion criteria: a histological diagnosis of prostate cancer, and after treatment of the primary disease, a diagnosis of biochemical relapse and no metastases or oligometastatic stage (less than 5 lesions) in conventional diagnostic images (bone scintigraphy, chest-abdominal and pelvic CT and pelvic MRI).
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
effectiveness of whole-body diffusion-weighted magnetic resonance imaging (WB-DW- MRI) in detecting metastases | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J Conde Moreno, MD PhD, Principal Investigator — Hospital Provincial de Castellon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conde-Moreno AJ, Herrando-Parreno G, Muelas-Soria R, Ferrer-Rebolleda J, Broseta-Torres R, Cozar-Santiago MP, Garcia-Pinon F, Ferrer-Albiach C. Whole-body diffusion-weighted magnetic resonance imaging (WB-DW-MRI) vs choline-positron emission tomography-computed tomography (choline-PET/CT) for selecting treatments in recurrent prostate cancer. Clin Transl Oncol. 2017 May;19(5):553-561. doi: 10.1007/s12094-016-1563-4. Epub 2016 Oct 31. PMID 27796820